CLINICAL TRIAL: NCT05706714
Title: Th1, Th2, Th17 Phenotype in Urea Cycle Disorders
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayca Kiykim, Associate Professor, Istanbul University - Cerrahpasa
Other Study IDs: IFUCD
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Urea Cycle Disorder; Lysinuric Protein Intolerance
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Lysinuric Protein Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with urea cycle disorder: Patients with inborn errors of metabolism resulting from defects in one of the enzymes or transporter molecules involved in the hepatic removal of ammonia from the bloodstream
- Patients with lysinuric protein intolerance: Patients with disorder caused by the body's inability to digest and use certain protein building blocks (amino acids), namely lysine, arginine, and ornithine
- Healthy control: Children without any comorbidity and chronic diseases.

SUMMARY:
Infection-related hyperammonemia in patients with urea cycle disorders is an important cause of morbidity and mortality. The relationship between immune system cells and the metabolic pathways used by these cells and inborn errors of metabolism is still under investigation. Current studies are generally based on experiments in mice. The investigators' goal is to study specific T cell subsets to understand the effects of the urea cycle on T cells.

The investigators collected blood samples from participants with lysinuric protein intolerance and urea cycle disorders for basic immunophenotyping, lymphocyte proliferation in response to phytohemagglutinin and CDmix, and cytokine analysis involving Th1, Th2, and Th17 and compared them with age-matched healthy controls. They also examined amino acid profiles in sera and supernatants before and after stimulation with PMA-ionomycin.

DETAILED DESCRIPTION:
The investigators aim to compare cellular immune response of T cell phenotype and proliferative functions in addition to lymphocyte subset analysis between urea cycle disorders and healthy controls.

Complete blood counts, immunoglobuline levels, lymptocyte subset analysis and Thelper cells will be analyzed. Additionally, T helper cells will be measured regarding their cytokine profile as Th1, Th2 and Th17. T cell proliferation response and aminoacid profiles in supernatants before and after stimulation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Children without any chronic conditions and having normal immunoglobulins and lymphocyte subsets

Exclusion Criteria:

* For healthy control, children having any signs for primary immune deficiencies

Max Age: 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with a diagnosis of urea cycle disorders and lysinuric protein intolerance
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Th1, Th2 and Th17 cells | baseline
  Th1, Th2 and Th17 cells will be measured following stimulation in cell culture

SECONDARY OUTCOMES:
Measurement of T cell proliferative capacity | baseline
  T cells' proliferation will be measured following stimulation in cell culture

OTHER OUTCOMES:
Measurement of amino acid profile changes before and after stimulation | baseline
  Serum Aminoacids from periphery, in cell culture supernatants before and after stimulation will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Kiykim, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)